CLINICAL TRIAL: NCT00860262
Title: An 8-week Randomised, Double-blind Study to Compare the Fixed-dose Combination of Telmisartan 80 mg & Amlodipine 10mg Versus Telmisartan 80 mg Monotherapy or Amlodipine 10 mg Monotherapy as First Line Therapy in Patients With Severe Hypertension (Grade 3).
Brief Title: Telmisartan and Amlodipine Fixed Dose Combination [FDC] Trial for the Treatment of Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.20; 2008-000873-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Telmisartan; telmisartan amlodipine combination

ARMS (3):
- telmisartan and amlodipine (Experimental): telmisartan and amlodipine used in combination vs amlodipine or telmisartan
  Interventions: Drug: telmisartan and amlodipine
- amlodipine (Active Comparator): telmisartan and amlodipine used in combination vs amlodipine or telmisartan
  Interventions: Drug: amlodipine
- telmisartan (Active Comparator): telmisartan and amlodipine used in combination vs amlodipine or telmisartan
  Interventions: Drug: telmisartan

INTERVENTIONS:
Drug: amlodipine — amlodipine 5mg for the first 2w then force titration to Amlodipine 10mg for remaining 6 w
  Arms: amlodipine
Drug: telmisartan — telmisartan 80mg for the 8w, no titration required
  Arms: telmisartan
Drug: telmisartan and amlodipine — telmisartan 80 and amlodipine 5mg for the first 2 weeks, then force titrated to telmisartan 80mg and amlodipine 10mg for the remaining 6w
  Arms: telmisartan and amlodipine

SUMMARY:
The primary objective of this trial is to demonstrate that following eight weeks of treatment the FDC of telmisartan 80 mg plus amlodipine 10 mg (T80/A10) is superior as first line therapy in reducing mean seated trough cuff Systolic Blood Pressure [SBP] compared to the monotherapies of telmisartan 80 mg (T80) and amlodipine 10 mg (A10) in patients with severe hypertension. A key secondary objective is to identify the duration of treatment required to demonstrate the superiority of the FDC over both of the monotherapies.

ELIGIBILITY:
Inclusion criteria

1. Ability to provide written informed consent in accordance with Good Clinical Practice and local legislation
2. Age 18 years or older
3. Patients with severe hypertension as defined SBP greater than 180 mmHg and DBP greater than 95 mmHg at randomisation
4. Ability to stop any current antihypertensive therapy without unacceptable risk to the patient (Investigators discretion)

Exclusion criteria Mean in-clinic seated cuff SBP >/= 200 mmHg and/or Diastolic Blood Pressure [DBP] >/= 95 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (137):
- United States (30):
  - 1235.20.525 Boehringer Ingelheim Investigational Site, Buena Park, California
  - 1235.20.503 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1235.20.507 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1235.20.529 Boehringer Ingelheim Investigational Site, Roseville, California
  - 1235.20.518 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1235.20.521 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 1235.20.508 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1235.20.506 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1235.20.519 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1235.20.523 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1235.20.528 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1235.20.516 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1235.20.527 Boehringer Ingelheim Investigational Site, Bay City, Michigan
  - 1235.20.510 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1235.20.512 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1235.20.509 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1235.20.511 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1235.20.515 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1235.20.534 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1235.20.526 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1235.20.513 Boehringer Ingelheim Investigational Site, Tipton, Pennsylvania
  - 1235.20.517 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 1235.20.522 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 1235.20.520 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1235.20.530 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1235.20.535 Boehringer Ingelheim Investigational Site, Draper, Utah
  - 1235.20.533 Boehringer Ingelheim Investigational Site, Magna, Utah
  - 1235.20.505 Boehringer Ingelheim Investigational Site, Saratoga Springs, Utah
  - 1235.20.537 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1235.20.501 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
- Bulgaria (9):
  - 1235.20.001 Boehringer Ingelheim Investigational Site, Burgas
  - 1235.20.002 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.003 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.005 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.006 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.007 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.008 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.009 Boehringer Ingelheim Investigational Site, Sofia
  - 1235.20.004 Boehringer Ingelheim Investigational Site, Stara Zagora
- Czechia (8):
  - 1235.20.052 Boehringer Ingelheim Investigational Site, Benátky nad Jizerou
  - 1235.20.059 Boehringer Ingelheim Investigational Site, Český Krumlov
  - 1235.20.051 Boehringer Ingelheim Investigational Site, Pilsen
  - 1235.20.053 Boehringer Ingelheim Investigational Site, Prague
  - 1235.20.054 Boehringer Ingelheim Investigational Site, Příbram
  - 1235.20.055 Boehringer Ingelheim Investigational Site, Slaný
  - 1235.20.057 Boehringer Ingelheim Investigational Site, Strakonice
  - 1235.20.058 Boehringer Ingelheim Investigational Site, Tábor
- France (32):
  - 1235.20.101A Boehringer Ingelheim Investigational Site, Albens
  - 1235.20.102F Boehringer Ingelheim Investigational Site, Arles
  - 1235.20.103A Boehringer Ingelheim Investigational Site, Béziers
  - 1235.20.103C Boehringer Ingelheim Investigational Site, Béziers
  - 1235.20.103F Boehringer Ingelheim Investigational Site, Béziers
  - 1235.20.106A Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1235.20.109B Boehringer Ingelheim Investigational Site, Brivé
  - 1235.20.108E Boehringer Ingelheim Investigational Site, Carbonne
  - 1235.20.101D Boehringer Ingelheim Investigational Site, Chambéry
  - 1235.20.103E Boehringer Ingelheim Investigational Site, Cournonterral
  - 1235.20.108C Boehringer Ingelheim Investigational Site, Cugnaux
  - 1235.20.106D Boehringer Ingelheim Investigational Site, Étrelles
  - 1235.20.108F Boehringer Ingelheim Investigational Site, Fenouillet
  - 1235.20.102A Boehringer Ingelheim Investigational Site, Gémenos
  - 1235.20.102C Boehringer Ingelheim Investigational Site, Gémenos
  - 1235.20.101C Boehringer Ingelheim Investigational Site, Grésy-sur-Aix
  - 1235.20.108A Boehringer Ingelheim Investigational Site, Labarthe-sur-Lèze
  - 1235.20.108B Boehringer Ingelheim Investigational Site, Labarthe-sur-Lèze
  - 1235.20.106F Boehringer Ingelheim Investigational Site, Louvigné-de-Bais
  - 1235.20.102E Boehringer Ingelheim Investigational Site, Marseille
  - 1235.20.106B Boehringer Ingelheim Investigational Site, Mordelles
  - 1235.20.107A Boehringer Ingelheim Investigational Site, Orthez
  - 1235.20.107B Boehringer Ingelheim Investigational Site, Orthez
  - 1235.20.107E Boehringer Ingelheim Investigational Site, Orthez
  - 1235.20.107G Boehringer Ingelheim Investigational Site, Orthez
  - 1235.20.109A Boehringer Ingelheim Investigational Site, Rosiers-d'Égletons
  - 1235.20.109F Boehringer Ingelheim Investigational Site, Saint-Aulaire
  - 1235.20.104A Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1235.20.104D Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1235.20.107F Boehringer Ingelheim Investigational Site, Salies-de-Béarn
  - 1235.20.105A Boehringer Ingelheim Investigational Site, Toulon
  - 1235.20.105D Boehringer Ingelheim Investigational Site, Toulon
- Hungary (9):
  - 1235.20.152 Boehringer Ingelheim Investigational Site, Budapest
  - 1235.20.156 Boehringer Ingelheim Investigational Site, Budapest
  - 1235.20.158 Boehringer Ingelheim Investigational Site, Budapest
  - 1235.20.159 Boehringer Ingelheim Investigational Site, Budapest
  - 1235.20.161 Boehringer Ingelheim Investigational Site, Budapest
  - 1235.20.153 Boehringer Ingelheim Investigational Site, Gyöngyös
  - 1235.20.154 Boehringer Ingelheim Investigational Site, Miskolc
  - 1235.20.157 Boehringer Ingelheim Investigational Site, Miskolc
  - 1235.20.155 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
- Romania (9):
  - 1235.20.252 Boehringer Ingelheim Investigational Site, Brăila
  - 1235.20.259 Boehringer Ingelheim Investigational Site, Bucharest
  - 1235.20.262 Boehringer Ingelheim Investigational Site, Bucharest
  - 1235.20.254 Boehringer Ingelheim Investigational Site, Iași
  - 1235.20.261 Boehringer Ingelheim Investigational Site, Oradea
  - 1235.20.256 Boehringer Ingelheim Investigational Site, Sibiu
  - 1235.20.251 Boehringer Ingelheim Investigational Site, Târgu Mureş
  - 1235.20.260 Boehringer Ingelheim Investigational Site, Tg. Mures
  - 1235.20.253 Boehringer Ingelheim Investigational Site, Timișoara
- Russia (11):
  - 1235.20.301 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.20.302 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.20.303 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.20.304 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.20.310 Boehringer Ingelheim Investigational Site, Moscow
  - 1235.20.305 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.20.306 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.20.307 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.20.308 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.20.309 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1235.20.311 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (6):
  - 1235.20.355 Boehringer Ingelheim Investigational Site, Galanta
  - 1235.20.353 Boehringer Ingelheim Investigational Site, Košice
  - 1235.20.352 Boehringer Ingelheim Investigational Site, Považská Bystrica
  - 1235.20.354 Boehringer Ingelheim Investigational Site, Rimavská Sobota
  - 1235.20.356 Boehringer Ingelheim Investigational Site, Trnava
  - 1235.20.351 Boehringer Ingelheim Investigational Site, Vráble
- South Korea (7):
  - 1235.20.207 Boehringer Ingelheim Investigational Site, Busan
  - 1235.20.206 Boehringer Ingelheim Investigational Site, Junam
  - 1235.20.205 Boehringer Ingelheim Investigational Site, Koyang
  - 1235.20.201 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.20.202 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.20.203 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.20.204 Boehringer Ingelheim Investigational Site, Seoul
- Spain (5):
  - 1235.20.406 Boehringer Ingelheim Investigational Site, Barcelona
  - 1235.20.408 Boehringer Ingelheim Investigational Site, Barcelona
  - 1235.20.402 Boehringer Ingelheim Investigational Site, Granada
  - 1235.20.403 Boehringer Ingelheim Investigational Site, Seville
  - 1235.20.409 Boehringer Ingelheim Investigational Site, Valencia
- Ukraine (11):
  - 1235.20.451 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.20.458 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.20.460 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1235.20.453 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.454 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.455 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.456 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.457 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.461 Boehringer Ingelheim Investigational Site, Kiev
  - 1235.20.452 Boehringer Ingelheim Investigational Site, Lviv
  - 1235.20.459 Boehringer Ingelheim Investigational Site, Odesa

RESULTS

PARTICIPANT FLOW:
Groups:
- T80+A10: Telmisartan 80 mg plus Amlodipine 10 mg once daily (T80+A10)
- Telmisartan 80 mg: Telmisartan 80 mg once daily (T80)
- Amlodipine 10 mg: Amlodipine 10 mg once daily (A10)
Period: Overall Study
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Started | 421 | 217 | 220
Completed | 401 | 195 | 202
Not Completed | 20 | 22 | 18
Not completed — Adverse Event | 9 | 6 | 7
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 8 | 6
Not completed — Lack of Efficacy | 0 | 4 | 3
Not completed — Other | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 421 | 217 | 220 | 858
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.4) | 58.1 (10.2) | 58.6 (10.5) | 58.2 (10.3)
Age, Customized [Number; unit: Participants]
  < 65 years | 309 | 158 | 156 | 623
  >= 65 years | 112 | 59 | 64 | 235
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 109 | 102 | 413
  Male | 219 | 108 | 118 | 445
Race/Ethnicity, Customized [Number; unit: participants]
  White | 362 | 186 | 190 | 738
  Black/African American | 34 | 15 | 15 | 64
  Asian | 20 | 14 | 14 | 48
  American Indian/Alaska Native | 5 | 1 | 0 | 6
  Hawaiian/Pacific Islander | 0 | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter] | 30.6 (5.9) | 30.2 (5.2) | 30.7 (6.3) | 30.6 (5.8)
Body Mass Index Class [Number; unit: participants]
  BMI < 25 | 63 | 31 | 35 | 129
  25 <= BMI < 30 | 160 | 79 | 82 | 321
  BMI >= 30 | 198 | 107 | 103 | 408
Race Class [Number; unit: participants]
  Non-Black | 387 | 202 | 205 | 794
  Black | 34 | 15 | 15 | 64
Type II Diabetes [Number; unit: participants]
  No | 349 | 183 | 197 | 729
  Yes | 72 | 34 | 23 | 129
Duration of Hypertension [Mean (Standard Deviation); unit: years] | 10.3 (9.6) | 9.4 (9.2) | 10.3 (10.1) | 10.1 (9.6)
Duration of Hypertension Class [Number; unit: participants]
  < 1 year | 38 | 25 | 20 | 83
  1 - 5 years | 124 | 64 | 72 | 260
  6 - 10 years | 103 | 61 | 54 | 218
  > 10 years | 156 | 67 | 74 | 297
Number of previous antihypertensive treatments [Number; unit: participants]
  0 | 49 | 37 | 26 | 112
  1 | 133 | 67 | 78 | 278
  2 | 136 | 59 | 71 | 266
  >= 3 | 103 | 54 | 45 | 202

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure (SBP) at Week 8
Description: Overall mean reduction from a common mean baseline in SBP
Time Frame: baseline and week 8
Population: Full analysis set (FAS) included all randomised patients who had at least one seated trough cuff SBP following administration of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 379 | 189 | 195
mmHg (millimeters of mercury) | -47.5 (0.69) | -36.9 (0.96) | -43.2 (0.95)
Statistical Analysis 1: Comparison: T80+A10 vs Telmisartan 80 mg; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -10.6, 95% CI 2-sided [-12.9 to -8.3], Standard Error of Mean 1.18 — Difference calculated as T80+A10 minus Telmisartan 80 mg
Statistical Analysis 2: Comparison: T80+A10 vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0002, Repeated measures ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-6.7 to -2.1], Standard Error of Mean 1.18 — Difference calculated as T80+A10 minus amlodipine 10 mg

2. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure at Week 6
Description: Overall mean reduction from a common mean baseline in SBP
Time Frame: baseline and week 6
Population: Full analysis set (FAS) included all patients who had efficacy data consisting of a baseline and at least one post-baseline trough BP measurement.
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 390 | 197 | 201
mmHg (millimeters of mercury) | -46.9 (0.73) | -36.3 (1.01) | -42.1 (1.01)
Statistical Analysis 1: Comparison: T80+A10 vs Telmisartan 80 mg; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -10.6, 95% CI 2-sided [-13.1 to -8.2], Standard Error of Mean 1.25 — Difference calculated as T80+A10 minus telmisartan 80 mg
Statistical Analysis 2: Comparison: T80+A10 vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-7.3 to -2.4], Standard Error of Mean 1.24 — Difference calculated as T80+A10 minus amlodipine 10 mg

3. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure at Week 4
Description: Overall mean reduction from a common mean baseline in SBP
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 202 | 203
mmHg (millimeters of mercury) | -44.5 (0.73) | -34.4 (1.01) | -39.8 (1.01)
Statistical Analysis 1: Comparison: T80+A10 vs Telmisartan 80 mg; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-12.6 to -7.7], Standard Error of Mean 1.24 — Difference calculated as T80+A10 minus telmisartan 80 mg
Statistical Analysis 2: Comparison: T80+A10 vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-7.2 to -2.4], Standard Error of Mean 1.24 — Difference calculated as T80+A10 minus amlodipine 10 mg

4. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure at Week 2
Description: Overall mean reduction from a common mean baseline in SBP
Time Frame: baseline and week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Groups:
- T80+A5: Telmisartan 80 mg plus Amlodipine 5 mg once daily (T80+A5)
- Amlodipine 5 mg: Amlodipine 5 mg once daily (A5)
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 395 | 208 | 204
mmHg (millimeters of mercury) | -37.9 (0.71) | -30.1 (0.97) | -33.3 (0.98)
Statistical Analysis 1: Comparison: T80+A5 vs Telmisartan 80 mg; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -7.8, 95% CI 2-sided [-10.2 to -5.4], Standard Error of Mean 1.20 — Difference calculated as T80+A10 minus telmisartan 80 mg
Statistical Analysis 2: Comparison: T80+A5 vs Amlodipine 5 mg; Test type: Superiority or Other; p = 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-7.0 to -2.3], Standard Error of Mean 1.21 — Difference calculated as T80+A10 minus amlodipine 10 mg

5. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure at Week 1
Description: Overall mean reduction from a common mean baseline in SBP
Time Frame: baseline and week 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
mmHg (millimeters of mercury) | -31.9 (0.72) | -25.4 (0.99) | -28.6 (0.99)
Statistical Analysis 1: Comparison: T80+A5 vs Telmisartan 80 mg; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-8.8 to -4.0], Standard Error of Mean 1.23 — Difference calculated as T80+A10 minus telmisartan 80 mg
Statistical Analysis 2: Comparison: T80+A5 vs Amlodipine 5 mg; Test type: Superiority or Other; p = 0.0077, Repeated measures ANCOVA; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-5.7 to -0.9], Standard Error of Mean 1.23 — Difference calculated as T80+A10 minus amlodipine 10 mg

6. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure (DBP) at Week 8
Description: Overall mean reduction from a common mean baseline in DBP
Time Frame: baseline and week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 379 | 189 | 195
mmHg (millimeters of mercury) | -18.7 (0.41) | -13.8 (0.58) | -16.3 (0.58)

7. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure at Week 6
Description: Overall mean reduction from a common mean baseline in DBP
Time Frame: baseline and week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 390 | 197 | 201
mmHg (millimeters of mercury) | -18.3 (0.41) | -13.5 (0.57) | -15.7 (0.57)

8. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure at Week 4
Description: Overall mean reduction from a common mean baseline in DBP
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 202 | 203
mmHg (millimeters of mercury) | -17.0 (0.43) | -12.1 (0.60) | -14.2 (0.60)

9. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure at Week 2
Description: Overall mean reduction from a common mean baseline in DBP
Time Frame: baseline and week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 395 | 208 | 204
mmHg (millimeters of mercury) | -13.2 (0.40) | -10.4 (0.56) | -11.4 (0.56)

10. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure at Week 1
Description: Overall mean reduction from a common mean baseline in DBP
Time Frame: baseline and week 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
mmHg (millimeters of mercury) | -10.9 (0.37) | -8.2 (0.50) | -9.6 (0.50)

11. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Control at Week 1
Description: Diastolic Blood Pressure Control is defined as achieving DBP < 90mmHg
Time Frame: week 1
Population: Full analysis set, imputation method used was last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
participants
  Controlled | 147 | 61 | 64
  Not Controlled | 240 | 146 | 143

12. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Control at Week 2
Description: DBP < 90 mmHg
Time Frame: week 2
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 405 | 212 | 212
participants
  Controlled | 205 | 87 | 91
  Not Controlled | 200 | 125 | 121

13. Secondary Outcome: Patients Achieving Blood Pressure Control at Week 1
Description: Blood Pressure Control is defined as achieving SBP< 140 mmHg and DBP < 90mmHg
Time Frame: week 1
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
participants
  Controlled | 54 | 16 | 15
  Not Controlled | 333 | 191 | 192

14. Secondary Outcome: Patients Achieving Blood Pressure Control at Week 2
Description: SBP < 140 mmHg and DBP < 90 mmHg
Time Frame: week 2
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 405 | 212 | 212
participants
  Controlled | 88 | 30 | 28
  Not Controlled | 317 | 182 | 184

15. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Response at Week 1
Description: Diastolic Blood Pressure Response is defined as achieving DBP < 90 mmHg or a reduction of >= 10 mmHg
Time Frame: baseline, week 1
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
participants
  Controlled | 232 | 95 | 100
  Not Controlled | 155 | 112 | 107

16. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Response at Week 2
Description: DBP < 90 mmHg or reduction of >= 10 mmHg
Time Frame: baseline, week 2
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 405 | 212 | 212
participants
  Controlled | 289 | 123 | 128
  Not Controlled | 116 | 89 | 84

17. Secondary Outcome: Patients Achieving Systolic Blood Pressure Response at Week 1
Description: Systolic Blood Pressure Response Control is defined as achieving SBP < 140 mmHg or a reduction of >= 15 mmHg
Time Frame: baseline, week 1
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
participants
  Controlled | 338 | 164 | 173
  Not Controlled | 49 | 43 | 34

18. Secondary Outcome: Patients Achieving Systolic Blood Pressure Response at Week 2
Description: SBP < 140 mmHg or reduction of >= 15 mmHg
Time Frame: baseline, week 2
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 405 | 212 | 212
participants
  Controlled | 387 | 169 | 189
  Not Controlled | 18 | 43 | 23

19. Secondary Outcome: Number of Patients Achieving Various Blood Pressure Response Levels at Week 1
Description: Optimal: SBP<120 and DBP< 80; Normal: 120<=SBP<130 and 80<= DBP<85; High normal: 130<=SBP<140 and 85<=DBP<90; High: SBP>=140 or DBP>=90
Time Frame: week 1
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 387 | 207 | 207
participants
  Optimal | 3 | 0 | 0
  Normal | 9 | 3 | 3
  High Normal | 42 | 13 | 12
  High | 333 | 191 | 192

20. Secondary Outcome: Number of Patients Achieving Various Blood Pressure Response Levels at Week 2
Description: as for outcome 19
Time Frame: week 2
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A5 | Telmisartan 80 mg | Amlodipine 5 mg
Number analyzed (Participants) | 405 | 212 | 212
participants
  Optimal | 6 | 0 | 0
  Normal | 21 | 7 | 5
  High Normal | 61 | 23 | 23
  High | 317 | 182 | 184

21. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Control at Week 4
Description: DBP < 90 mmHg
Time Frame: week 4
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 212 | 203
participants
  Controlled | 268 | 106 | 109
  Not Controlled | 124 | 106 | 94

22. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Control at Week 6
Description: DBP < 90 mmHg
Time Frame: week 6
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Controlled | 290 | 110 | 128
  Not Controlled | 104 | 102 | 77

23. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Control at Week 8
Description: DBP < 90 mmHg
Time Frame: week 8
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Controlled | 291 | 112 | 131
  Not Controlled | 103 | 100 | 74

24. Secondary Outcome: Patients Achieving Blood Pressure Control at Week 4
Description: SBP < 140 mmHg and DBP < 90 mmHg
Time Frame: week 4
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 212 | 203
participants
  Controlled | 161 | 49 | 53
  Not Controlled | 231 | 163 | 150

25. Secondary Outcome: Patients Achieving Blood Pressure Control at Week 6
Description: SBP < 140 mmHg and DBP < 90 mmHg
Time Frame: week 6
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Controlled | 196 | 54 | 77
  Not Controlled | 198 | 158 | 128

26. Secondary Outcome: Patients Achieving Blood Pressure Control at Week 8
Description: SBP < 140 mmHg and DBP < 90 mmHg
Time Frame: week 8
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 395 | 212 | 205
participants
  Controlled | 199 | 51 | 73
  Not Controlled | 196 | 161 | 132

27. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Response at Week 4
Description: DBP < 90 mmHg or reduction of >= 10 mmHg
Time Frame: baseline, week 4
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 212 | 212
participants
  Controlled | 339 | 132 | 151
  Not Controlled | 53 | 80 | 61

28. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Response at Week 6
Description: DBP < 90 mmHg or reduction of >= 10 mmHg
Time Frame: baseline, week 6
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Controlled | 356 | 144 | 168
  Not Controlled | 38 | 68 | 37

29. Secondary Outcome: Patients Achieving Diastolic Blood Pressure Response at Week 8
Description: DBP < 90 mmHg or reduction of >= 10 mmHg
Time Frame: baseline, week 8
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 395 | 212 | 205
participants
  Controlled | 361 | 147 | 172
  Not Controlled | 34 | 65 | 33

30. Secondary Outcome: Patients Achieving Systolic Blood Pressure Response at Week 4
Description: SBP < 140 mmHg or reduction of >= 15 mmHg
Time Frame: baseline, week 4
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 212 | 203
participants
  Controlled | 388 | 180 | 194
  Not Controlled | 4 | 32 | 9

31. Secondary Outcome: Patients Achieving Systolic Blood Pressure Response at Week 6
Description: SBP < 140 mmHg or reduction of >= 15 mmHg
Time Frame: baseline, week 6
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Controlled | 388 | 184 | 201
  Not Controlled | 6 | 28 | 4

32. Secondary Outcome: Patients Achieving Systolic Blood Pressure Response at Week 8
Description: SBP < 140 mmHg or reduction of >= 15 mmHg
Time Frame: baseline, week 8
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 395 | 212 | 205
participants
  Controlled | 391 | 188 | 202
  Not Controlled | 4 | 24 | 3

33. Secondary Outcome: Patients Achieving Normal Blood Pressure Response at Week 4
Description: as for outcome 19
Time Frame: week 4
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 392 | 212 | 203
participants
  Optimal | 15 | 4 | 2
  Normal | 47 | 15 | 14
  High Normal | 99 | 30 | 37
  High | 231 | 163 | 150

34. Secondary Outcome: Patients Achieving Normal Blood Pressure Response at Week 6
Description: as for outcome 19
Time Frame: week 6
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 394 | 212 | 205
participants
  Optimal | 17 | 5 | 3
  Normal | 73 | 19 | 18
  High Normal | 106 | 30 | 56
  High | 198 | 158 | 128

35. Secondary Outcome: Patients Achieving Normal Blood Pressure Response at Week 8
Description: as for outcome 19
Time Frame: week 8
Population: FAS (LOCF)
Measure: Number; unit: participants
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Number analyzed (Participants) | 395 | 212 | 205
participants
  Optimal | 18 | 3 | 2
  Normal | 76 | 21 | 25
  High Normal | 105 | 27 | 46
  High | 196 | 161 | 132

ADVERSE EVENTS:
Time Frame: First study medication intake, last study medication intake + 6 days
Arm/Group | T80+A10 | Telmisartan 80 mg | Amlodipine 10 mg
Serious Adverse Events (participants affected / at risk) | 3/421 | 2/217 | 2/220
Other Adverse Events (participants affected / at risk) | 67/421 | 25/217 | 42/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T80+A10 (N=421) | Telmisartan 80 mg (N=217) | Amlodipine 10 mg (N=220)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T80+A10 (N=421) | Telmisartan 80 mg (N=217) | Amlodipine 10 mg (N=220)
Oedema peripheral (General disorders) | 55 | 8 | 33
Headache (Nervous system disorders) | 16 | 18 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.